CLINICAL TRIAL: NCT00001992
Title: A Phase I Study of the Safety and Immunogenicity of Rgp 120/HIV-1IIIB Vaccine in HIV-1 Seropositive Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Prevention
Other Study IDs: 075A; V0200g
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-08

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS Vaccines
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Biological: rgp120/HIV-1IIIB

SUMMARY:
To test the safety and immunogenicity of rgp 120/HIV-1IIIB vaccine in HIV-1 seropositive adult patients.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Stage 1 or 2 Walter Reed clinical staging of HIV infected individuals.
* The ability to understand and sign a written informed consent form, which must be obtained prior to study entry.
* Be available for 24 weeks so that follow up may be completed.
* Qualify for care as Department of Defense health care beneficiary.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Prior history of clinically significant cardiac, pulmonary, hepatic, renal, neurologic or autoimmune disease, other than HIV-1 infection, and in less than average general health as determined by a medical history, physical examination, and the required laboratory test results.

Concurrent Medication:

Excluded:

* Corticosteroids or other known immunosuppressive drugs.
* Any experimental agents.

Patients with the following are excluded:

* Prior history of clinically significant cardiac, pulmonary, hepatic, renal, neurologic or autoimmune disease, other than HIV-1 infection, and in less than average general health as determined by a medical history, physical examination, and the required laboratory test results.

Prior Medication:

Excluded within 30 days of study entry:

* Zidovudine or other anti-retroviral agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed Army Institute of Research, Rockville, Maryland, United States